CLINICAL TRIAL: NCT00332852
Title: An Open Phase III Trial With Letrozole as Early Adjuvant Treatment of Postmenopausal Patients With Primary Breast Cancer
Brief Title: Letrozole as Early Adjuvant Treatment of Postmenopausal Patients With Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345DDE10
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Postive breast cancer; postmenopausal; disease free survival; letrozole; early adjuvant treatment; primary hormone receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — 2.5 mg/day - oraly
  Other Names: Femara; FEM345

SUMMARY:
This is a prospective open-label one-arm phase III trial designed to evaluate the safety and efficacy of letrozole 2.5 mg administered orally daily for 24 months as adjuvant therapy in postmenopausal patients with primary breast cancer.

This trial is not recruiting patients in the United States.

ELIGIBILITY:
Inclusion criteria:

* Compliant postmenopausal women with primary operable breast cancer after complete surgery and suitable for endocrine treatment
* Nodal status negative or positive
* Good Health status 0-2 (Eastern Cooperative Oncology Group)
* Estrogen- and/or progesterone-receptor positive
* Adequate marrow, kidney and liver function

Exclusion criteria:

* Metastatic or inflammatory breast cancer
* Patients with previous or concomitant cancers (not breast cancer) within the past 5 years EXCEPT adequately treated basal or squamous cell skin cancer or in situ cancer of the cervix. Patients with other previous cancers must have been disease-free for at least 5 years and Patients with uncontrolled, non-malignant systemic cardiovascular, kidney, and liver diseases.
* Current/active dental problems including infection of the teeth or jawbone, dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw, of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery
* Patients with primary overactive parathyroid
* Patients with a known hypersensitivity to zoledronic acid or other bisphosphonates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients without recurrence after 24 months of Letrozole treatment as assessed by radiological imaging | after 24 months

SECONDARY OUTCOMES:
Disease free survival (DFS) | every 6 months for 24 months
Quality of life as assessed by EORTC QLQ-C30 + BR23 every 3 months | Every 6 months
Safety and tolerability with assessments incuding biochemistry, hematology, ECG, pyhsical exam and AE documentation | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (53):
- Germany (53):
  - Novartis Investigative Site, Albstadt
  - Schorndorf, Augsburg
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Holzminden
  - Novartis Investigative Site, Höxter
  - Novartis Investigative Site, Ilsede
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Konigs
  - Schorndorf, Konstanz
  - Novartis Investigative Site, Lich
  - Novartis Investigative Site, Lohsa/Weisskollm
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Saint Wendel
  - Novartis Investigative Site, Salzgitter
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwetzingen
  - Novartis Investigative Site, Starnberg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tuttlingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Walsrode
  - Novartis Investigative Site, Westerburg
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wolfsburg